CLINICAL TRIAL: NCT07053839
Title: Effect of the Visual Reminder "AdhasText" on Adherence to Inhaled Corticosteroids, Symptom Control, and Pulmonary Function in Children With Asthma: A Randomized Clinical Trial
Brief Title: Effect of a Daily Text Reminder on Asthma Medication Use, Symptom Control, and Lung Function in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ROXANA AZNARAN TORRES (Other)
Responsible Party: Sponsor-Investigator, ROXANA AZNARAN TORRES, Principal investigator, MD, PhD, Universidad Privada Antenor Orrego
Organization: Universidad Privada Antenor Orrego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0726-2023-UPAO; 0422-2023-D-EPG-UPAO (Other: Universidad Privada Antenor Orrego Graduate School)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Asthma in Children
Keywords: Text message; asthma; treatment adherence; symptom control; spirometry; children
MeSH Terms: conditions — Asthma; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Text Reminder (AdhasText) (Experimental): Participants in this group will receive a daily text message reminder ("AdhasText") to encourage them to use their inhalers regularly for 90 days. They will continue with their regular asthma management as prescribed by their healthcare providers.
  Interventions: Behavioral: Daily Text Reminder
- Usual care (No Intervention): Participants in this group will receive the usual care for asthma, which does not include the daily text message reminders. They will continue with their regular asthma management as prescribed by their healthcare providers.

INTERVENTIONS:
Behavioral: Daily Text Reminder — The intervention, titled "AdhasText," involved sending a daily SMS reminder to caregivers, specifically mothers of children with asthma. The message, "If you want to stay healthy, you must use your inhaler," was sent at 7:00 p.m. over a 90 days period.
  Arms: Daily Text Reminder (AdhasText)

SUMMARY:
The goal of this clinical trial is to learn if a daily text reminder ("AdhasText") can help children with asthma use their inhalers regularly, control their symptoms, and improve their lung function. The main questions it aims to answer are:

Does the daily text reminder improve adherence to inhaled corticosteroids in children with asthma? Does the text reminder help children with asthma control their symptoms better? Does the text reminder improve lung function in children with asthma?

Researchers will compare children who receive the daily text reminder with usual care to children who receive usual care (without the reminder) to see if the text reminder improves adherence, symptom control, and lung function.

Participants will:

Receive a daily text reminder or usual care (no reminder) for 90 days Complete questionnaires about their asthma symptoms at 45 and 90 days Have spirometry tests to measure lung function at the start of the study and 90 days

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 14 years with a clinical diagnosis of asthma
* Children who required initiation of treatment with a fixed and regular dose of inhaled corticosteroids
* Mothers or caregivers who had a mobile phone capable of sending and receiving text messages

Exclusion Criteria:

* Children with congenital heart disease
* Children who were unable to perform baseline spirometry
* Children who experienced at least one exacerbation during the pre-randomization period

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Inhaler Adherence as Measured by the Inhaler Adherence Scale for Children (IASC) at 45 and 90 Days | 45 days (T1) and 90 days (T2) after the intervention
  Inhaler adherence was measured using the Inhaler Adherence Scale for Children (IASC), which evaluates adherence across three domains: Cognitive, Psychosocial, and Control & Autonomy. The scale consists of 12 questions, with responses ranging from 0 (indicating poor adherence) to 4 (indicating full adherence) for each question. A higher total score indicates better adherence.

SECONDARY OUTCOMES:
Change in Asthma Symptom Control as Measured by the ACT (Asthma Control Test) and c-ACT (Childhood Asthma Control Test) at 45 and 90 Days | Day 45 and day 90 after the intervention
  Symptom control was assessed using the Asthma Control Test (ACT) for participants aged 12 years and older, and the Childhood Asthma Control Test (c-ACT) for children under 12 years old. The ACT consists of 5 questions regarding asthma symptoms, and the c-ACT includes 4 questions for the child and 3 for the caregiver. A higher score indicates better control over asthma symptoms.
Change in Pulmonary Function as Measured by Spirometry at 90 Days | Baseline and day 90 after the intervention
  Pulmonary function was assessed using spirometry at 90 days (T2). This measure evaluates the participants' lung function by assessing key parameters such as Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC). A bronchodilator response (BDR) was defined as an increase of more than 10% in FEV₁ or FVC following the administration of 400 µg of inhaled salbutamol; responses below this threshold indicated absence of BDR. Pulmonary function was categorized into four groups: (1) normal baseline spirometry without BDR (considered the only normal pattern), (2) normal baseline spirometry with BDR, (3) obstructive pattern without BDR, and (4) obstructive pattern with BDR. Additionally, lung function impairment severity was classified using z-score values: > -1.645 (normal), -1.65 to -2.5 (mild), -2.51 to -4 (moderate), and < -4.1 (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Docente de Trujillo, Trujillo, La Libertad, Peru

IPD SHARING:
Plan to Share IPD: No
The informed consent signed by participants does not include authorization to share individual-level data with external researchers.

REFERENCES:
- [Background] Jeminiwa R, Hohmann L, Qian J, Garza K, Hansen R, Fox BI. Impact of eHealth on medication adherence among patients with asthma: A systematic review and meta-analysis. Respir Med. 2019 Mar;149:59-68. doi: 10.1016/j.rmed.2019.02.011. Epub 2019 Feb 15. PMID 30803887
- [Background] Chan AH, Stewart AW, Harrison J, Camargo CA Jr, Black PN, Mitchell EA. The effect of an electronic monitoring device with audiovisual reminder function on adherence to inhaled corticosteroids and school attendance in children with asthma: a randomised controlled trial. Lancet Respir Med. 2015 Mar;3(3):210-9. doi: 10.1016/S2213-2600(15)00008-9. Epub 2015 Jan 21. PMID 25617215
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Morton RW, Everard ML, Elphick HE. Adherence in childhood asthma: the elephant in the room. Arch Dis Child. 2014 Oct;99(10):949-53. doi: 10.1136/archdischild-2014-306243. Epub 2014 May 29. PMID 24876303
- [Background] Papi A, Brightling C, Pedersen SE, Reddel HK. Asthma. Lancet. 2018 Feb 24;391(10122):783-800. doi: 10.1016/S0140-6736(17)33311-1. Epub 2017 Dec 19. PMID 29273246